CLINICAL TRIAL: NCT04422418
Title: Multi-Center Prospective Cohort Study: Impact of Burnout on Cardiovascular and Immune Biomarkers Among Frontline Healthcare Professionals During Covid-19 Pandemic in Abu Dhabi Emirate
Brief Title: Impact of Burnout on Cardiovascular and Immune Biomarkers in Healthcare Professionals - Covid-19 Pandemic in Abu Dhabi
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Khalifa University for Science and Technology (Other)
Collaborators: Zayed Military Hospital (Other Government); Abu Dhabi University (Unknown); Cleveland Clinic Abu Dhabi (Other); Sheikh Khalifa Medical City (Other); Sheikh Shakhbout Medical City (Other); Mediclinic Middle East (Industry); Myriad Global Solutions (Unknown)
Responsible Party: Sponsor
Other Study IDs: CPRA-2020-034
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-06

CONDITIONS: Cardiovascular Risk Factor; Burnout; Immune Deficiency
Keywords: Pandemics; Healthcare professionals; Burnout; Cardiovascular risk
MeSH Terms: conditions — Burnout, Psychological; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of our project is to investigate the evolution of psychosocial, cardiovascular and immune markers in healthcare with different levels of exposure to the COVID-19 pandemic.

DETAILED DESCRIPTION:
Introduction: The coronavirus disease 2019 (COVID-19) pandemic has created new and unpredictable challenges for healthcare systems. Healthcare professionals are heavily affected by this rapidly changing situation. They may experience psychological burden, especially nurses, women, and frontline health care professionals directly engaged in the diagnosis, treatment, and care for patients with COVID-19. The objective of this study is to investigate the evolution of psychosocial, cardiovascular and immune markers in healthcare professionals with different levels of exposure to the COVID-19 pandemic. The effects of the pandemic work burden on psychological, cardiovascular and immune biomarkers will be stratified per level of exposure to the COVID-19 pandemic, positive diagnosis to COVID-19, profession, sex, age and already existent cardiovascular risk.

Methods: A STROBE compliant, blended exploratory study involving online and onsite approach with wearable monitoring will be implemented. A planned random probability sample of residents, staff physicians, nurses and auxiliary healthcare professionals will be recruited from both inpatient and outpatient medicine services will be stratified by exposure to COVID-19 pandemic (frontline versus second line). In a first step, will be an online recruitment with e-consent and e-survey with Maslach Burnout Inventory, Fuster-BEWAT score and sociodemographic characteristics, and planning for onsite visit; in a second step, will be a setup for wearable monitoring of heart rate, actimetry and sleep quality together with blood sampling for immune biomarkers; steps 1 & 2 will be repeated at 2-3 months, 6 months. Power BI & Tableau will be used for data visualization purposes, while the front-end data capture application will be used for data collection and will be built using specific survey/questionnaire related tools for healthcare usage data linkage.

Ethics and dissemination: Institutional Review Board approval has been obtained from Khalifa University (protocol # CPRA-2020-034) and Department of Health-Abu Dhabi (protocol # CVDC-20-05/2020-8). Data analysis, release of results and publication of manuscripts are scheduled to start in early 2021. Data and findings may be useful to healthcare policymakers for developing preventive strategies to reduce or prevent burnout, cardiovascular risk and immune dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* all residents, staff physicians, nurses and auxiliary healthcare professionals from both inpatient and outpatient medicine services who agreed to be a part of the study will be provided with heart rate tracking devices to monitor heart rate.

Exclusion Criteria:

* not willing to complete written consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents, staff physicians, nurses and auxiliary healthcare professionals (adult males and females over 18 years) from both inpatient and outpatient medicine services
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-14 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Burnout at 2-3 months and 6 months | baseline, 2-3 months, 6 months
  Burnout - through self-reported stress and burnout thoughts, beliefs, emotions, behavior related to Covid-19 using Maslach Burnout Inventory. Maslach Burnout Inventory - is a 22-item survey that covers 3 areas: Emotional Exhaustion (EE), Depersonalization (DP), and low sense of Personal Accomplishment (PA). Each subscale includes multiple questions with frequency rating choices of Never, A few times a year or less, Once a month or less, A few times a month, Once a week, A few times a week, or Every day.
Change from Baseline Cardiovascular Risk Cardiovascular Risk Through Heart Rate Variability Markers at 2-3 months and 6 months | baseline, 2-3 months, 6 months
  Data is collected through wearable monitoring technology. Cardiovascular risk through monitoring of heart rate variability (HRV) markers. Changes of heart rate variability (HRV) reflecting cardiac autonomic dysfunction are associated with greater risks for cardiac morbidity and mortality.
Change from Baseline Through Actigraphy at 2-3 months and 6 months | baseline, 2-3 months, 6 months
  Data is collected through wearable monitoring technology. Actigraphy data is collected in 1 min epochs using the zero-crossing modes.
Change from Baseline Through Sleep Quality at 2-3 months and 6 months | baseline, 2-3 months, 6 months
  Data is collected through wearable monitoring technology. Sleep efficiency is defined as the proportion of the estimated sleep periods spent asleep. Sleep latency is the length of time taken to fall asleep, calculated as the time between 'lights off' to the first period of 3 min of consecutive epochs scored as sleep.
Change from Baseline Cardiovascular Risk Through Fuster-BEWAT score at 2-3 months and 6 months | baseline, 2-3 months, 6 months
  Cardiovascular risk through Fuster-BEWAT score. The Fuster-BEWAT score will be analyzed as a continuous variable with total score ranging from 0 to 15 points. Additionally, each component will be categorized as ideal (3) or nonideal (0 to 2), and participants will be classified as having poor, intermediate, or ideal cardiovascular health based on the total number of ideal components (0 to 1 = poor, 2 to 3 = intermediate, 4 to 5 = ideal) (Fernández-Alvira et al., 2017).
Change from Baseline Immune Dysfunction at 2-3 months and 6 months | baseline, 2-3 months, 6 months
  Classification of the immune function will be screened.

SECONDARY OUTCOMES:
Change from Baseline Cardio-Respiratory Fitness at 2-3 months and 6 months | baseline, 2-3 months, 6 months
  Submaximal field test and maximal oxygen consumption (VO2, mL/kg/min).

CONTACTS AND LOCATIONS:
Overall Officials: Wael Almahmeed, MD, Study Chair — Cleveland Clinic Abu Dhabi
Locations (4):
- United Arab Emirates (4):
  - Cleveland Clinic Abu Dhabi, Abu Dhabi
  - Mediclinic, Abu Dhabi
  - Sheikh Khalifa Medical City, Abu Dhabi
  - Sheikh Shakhbout Medical City, Abu Dhabi

REFERENCES:
- [Background] Pereira VL Jr, Dobre M, Dos Santos SG, Fuzatti JS, Oliveira CR, Campos LA, Brateanu A, Baltatu OC. Association between Carotid Intima Media Thickness and Heart Rate Variability in Adults at Increased Cardiovascular Risk. Front Physiol. 2017 Apr 26;8:248. doi: 10.3389/fphys.2017.00248. eCollection 2017. PMID 28491040
- [Background] Pinheiro Ade O, Pereira VL Jr, Baltatu OC, Campos LA. Cardiac autonomic dysfunction in elderly women with myocardial infarction. Curr Med Res Opin. 2015;31(10):1849-54. doi: 10.1185/03007995.2015.1074065. Epub 2015 Aug 26. PMID 26196167
- [Background] da Silva ELP, Pereira R, Reis LN, Pereira VL Jr, Campos LA, Wessel N, Baltatu OC. Heart rate detrended fluctuation indexes as estimate of obstructive sleep apnea severity. Medicine (Baltimore). 2015 Jan;94(4):e516. doi: 10.1097/MD.0000000000000516. PMID 25634206
- [Background] Gomez-Pardo E, Fernandez-Alvira JM, Vilanova M, Haro D, Martinez R, Carvajal I, Carral V, Rodriguez C, de Miguel M, Bodega P, Santos-Beneit G, Penalvo JL, Marina I, Perez-Farinos N, Dal Re M, Villar C, Robledo T, Vedanthan R, Bansilal S, Fuster V. A Comprehensive Lifestyle Peer Group-Based Intervention on Cardiovascular Risk Factors: The Randomized Controlled Fifty-Fifty Program. J Am Coll Cardiol. 2016 Feb 9;67(5):476-85. doi: 10.1016/j.jacc.2015.10.033. Epub 2015 Nov 9. PMID 26562047
- [Background] Fernandez-Alvira JM, Fuster V, Pocock S, Sanz J, Fernandez-Friera L, Laclaustra M, Fernandez-Jimenez R, Mendiguren J, Fernandez-Ortiz A, Ibanez B, Bueno H. Predicting Subclinical Atherosclerosis in Low-Risk Individuals: Ideal Cardiovascular Health Score and Fuster-BEWAT Score. J Am Coll Cardiol. 2017 Nov 14;70(20):2463-2473. doi: 10.1016/j.jacc.2017.09.032. PMID 29145946
- [Background] Henriksen A, Grimsgaard S, Horsch A, Hartvigsen G, Hopstock L. Validity of the Polar M430 Activity Monitor in Free-Living Conditions: Validation Study. JMIR Form Res. 2019 Aug 16;3(3):e14438. doi: 10.2196/14438. PMID 31420958
- [Derived] Alameri F, Aldaheri N, Almesmari S, Basaloum M, Albeshr NA, Simsekler MCE, Ugwuoke NV, Dalkilinc M, Al Qubaisi M, Campos LA, Almahmeed W, Alefishat E, Al Tunaiji H, Baltatu OC. Burnout and Cardiovascular Risk in Healthcare Professionals During the COVID-19 Pandemic. Front Psychiatry. 2022 Apr 4;13:867233. doi: 10.3389/fpsyt.2022.867233. eCollection 2022. PMID 35444572
- [Derived] Al Tunaiji H, Al Qubaisi M, Dalkilinc M, Campos LA, Ugwuoke NV, Alefishat E, Aloum L, Ross R, Almahmeed W, Baltatu OC. Impact of COVID-19 Pandemic Burnout on Cardiovascular Risk in Healthcare Professionals Study Protocol: A Multicenter Exploratory Longitudinal Study. Front Med (Lausanne). 2020 Dec 22;7:571057. doi: 10.3389/fmed.2020.571057. eCollection 2020. PMID 33415114